CLINICAL TRIAL: NCT00635375
Title: A Comparative Study Between BiliSoft Blue LED Fiberoptic Blanket Phototherapy, Giraffe Spot PT Phototherapy, Natus Blue LED Bank Light Phototherapy, and BiliSoft + Giraffe Spot PT Combination Therapy
Brief Title: Comparative Study of Phototherapy for Hyperbilirubinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Lynn Lynam, MIC Clinical Programs & Research, GE Healthcare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8828882
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): LED fiberoptic blanket phototherapy
  Interventions: Device: LED fiberoptic blanket phototherapy (BiliSoft blue LED fiberoptic blanket phototherapy)
- 2 (Experimental): metal halide phototherapy
  Interventions: Device: Metal halide phototherapy (Spot PT metal halide phototherapy)
- 3 (Active Comparator): LED bank phototherapy
  Interventions: Device: LED bank phototherapy (Natus neoBlue LED bank phototherapy)
- 4 (Experimental): Combination metal halide phototherapy plus LED fiberoptic blanket phototherapy
  Interventions: Device: Metal halide plus LED fiberoptic blanket phototherapy (BiliSoft and Spot PT)

INTERVENTIONS:
Device: LED fiberoptic blanket phototherapy (BiliSoft blue LED fiberoptic blanket phototherapy) — 35-50 mW/cm2/nm
  Other Names: BiliSoft blue LED fiberoptic blanket phototherapy
  Arms: 1
Device: Metal halide phototherapy (Spot PT metal halide phototherapy) — 29.3-57.6 mW/cm2/nm
  Other Names: Spot PT metal halide phototherapy
  Arms: 2
Device: LED bank phototherapy (Natus neoBlue LED bank phototherapy) — 12-35 mW/cm2/nm
  Other Names: Natus neoBlue LED bank phototherapy
  Arms: 3
Device: Metal halide plus LED fiberoptic blanket phototherapy (BiliSoft and Spot PT) — 29.3-57.6 mW/cm2/nm and 35-50 mW/cm2/nm
  Other Names: BiliSoft and Spot PT
  Arms: 4

SUMMARY:
Hyperbilirubinemia is a common problem for term and preterm newborns in intensive care nurseries around the world. It is a condition in which there is too much bilirubin in the blood. Bilirubin is a substance that is naturally released when red blood cells break down. In the early newborn period, multiple factors lead to an abnormally elevated bilirubin level. Large amounts of bilirubin can circulate to tissues in the brain and may cause seizures or brain damage. About 6.1% of term newborns and a higher percentage of preterm newborns develop hyperbilirubinemia that requires treatment. Initiating treatment depends on many factors, including the cause of the hyperbilirubinemia, the level of serum indirect bilirubin, the rate of indirect bilirubin rise, and the age of the patient. The goal of treatment is to keep the level of bilirubin from rising to dangerous levels.

The bilirubin molecule absorbs light. Therefore, treatment of hyperbilirubinemia involves exposure of the baby's skin to special blue spectrum light. Phototherapy is globally recognized as the standard of care for treatment of elevated indirect hyperbilirubinemia in the neonatal period. This light exposure converts water-insoluble indirect bilirubin to a more easily excreted soluble molecule. Over the last five years, several devices have been introduced that emit high intensity light in the blue portion of the visible light spectrum. However, despite frequent use of such therapy, the effectiveness of different phototherapy devices has not been adequately compared. The objective of this study is to compare the efficacy of the blue LED fiberoptic phototherapy with the metal halide spot phototherapy versus blue LED bank light phototherapy versus a combination of tandem therapy on lowering to total serum bilirubin.

ELIGIBILITY:
Inclusion Criteria:

* > 23 0/7 weeks gestation
* > 500 grams
* Non-hemolytic or presumed physiologic jaundice (within the first 14 days of life)

Exclusion Criteria:

* Known congenital infection (proven bacterial or viral etiology)
* Known hemolytic diseases such as but not limited to ABO or Rh incompatibility, minor blood group incompatibility, glucose-6-phosphate dehydrogenase deficiency, or hereditary red blood cell membrane defects (Coombs or DAT positive)
* Suspected genetic, syndromic, or hepatic disorder-

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The LED Fiberoptic Phototherapy System and metal halide spot phototherapy are will show no difference in therapeutic treatment times compared to the LED Bank Light System. | 14 months

SECONDARY OUTCOMES:
Combination Phototherapy Systems will show a 20% shorter treatment time compared to single treatment methods alone. | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Sturtz, MD, Principal Investigator — Christiana Hospital
Locations (2):
- United States (2):
  - Christiana Hospital, Newark, Delaware
  - University of Tennessee, Knoxville, Tennessee